CLINICAL TRIAL: NCT02506101
Title: Randomized, Split-Body, Single-Blinded Clinical Trial of Narrow Band-Ultraviolet B (NB-UVB) Treatment for Vitiligo
Brief Title: Randomized, Split-body, Single-blinded Clinical Trial of NB-UVB Treatment for Vitiligo
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment and staff availability to administer treatment.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00052103
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Vitiligo; Pigmentation; Dyschromia
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- narrow-band ultraviolet B phototherapy (Experimental): We will use the 3 Series PC & SP Phototherapy Cabinet for treatment of vitiligo.
  Interventions: Device: narrow-band ultraviolet B phototherapy
- no intervention (No Intervention): untreated

INTERVENTIONS:
Device: narrow-band ultraviolet B phototherapy — There are two types of UVB: broad band and narrow band, with the major difference being that narrow band emits a smaller range of ultraviolet light, typically 311-312 nm. NB-UVB is a clinically indicated treatment for vitiligo lesions and treatments are usually administered in an outpatient setting 3 times a week.
  Arms: narrow-band ultraviolet B phototherapy

SUMMARY:
The objective of this study is to assess the effectiveness and safety of narrowband-ultraviolet B (NB-UVB) treatment in adult subjects with vitiligo.

DETAILED DESCRIPTION:
Vitiligo is a chronic acquired cutaneous disease of pigmentation that affects patients' quality of life across all degrees of involvement and severity. Phototherapy is a clinically indicated treatment for skin lesions. Treatments are usually administered in an outpatient setting, typically three times per week. This is a proof-of-concept study as there are few well-designed prospective clinical studies showing the efficacy of NB-UVB phototherapy in the treatment of vitiligo in terms of repigmentation and quality of life. The following are the proposed objectives of this study:

1. NB-UVB phototherapy improves vitiligo with at least 50% repigmentation compared to no treatment on affected areas of the trunk and extremities over 24 weeks.
2. NB-UVB phototherapy leads to improvement in quality of life as measured by standardized quality of life metrics (DLQI and Skindex-29) over 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older with bilateral symmetrical vitiligo lesions, in general good health as determined by the Principal Investigator by medical history and physical exam.
* Able to understand consent procedure
* Able to comply with protocol activities
* If a woman, before entry she must be:

  1. postmenopausal, defined as 45 years of age with amenorrhea for at least 18 months, or >45 years of age with amenorrhea for at least 6 months and a serum follicule stimulating hormone (FSH) level >40 IU/mL, or surgically postmenopausal (bilateral oophorectomy), or
  2. surgically sterile (have had a hysterectomy or tubal ligation or otherwise be incapable of pregnancy), or
  3. If heterosexually active and of childbearing potential, practicing a highly effective method of birth control, (examples include hormonal prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method (e.g. condoms, diaphragms, or cervical cap, with spermicidal foam, cream, or gel), or male partner sterilization consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials, for the duration of their participation in the study, or
  4. Not heterosexually active

Exclusion Criteria:

* Patients less than 18 years old
* Patients not able to understand consent procedure
* Patients unable to comply with protocol activities
* Patients that do not have bilateral symmetrical vitiligo lesions
* Non-English speakers: the study assessments/questionnaires/evaluations are not scientifically validated in languages other than English. Given the lack of translators in over 50% of patient encounters in the dermatology clinic and the interpreters' limited time commitments when one does show up, it is impossible to safely enroll or follow patients who do not speak English. Phone translators are impossible given that we have written consent forms, which often exceed 10 pages in length.
* Patients with a photosensitive disorder or on a medication which has been demonstrated in these patients to cause photosensitivity
* Patients receiving concomitant phototherapy to test sites
* Patient receiving topical medication to test sites within 2 weeks of study initiation
* Patient receiving oral medications for vitiligo within 4 weeks prior to study initiation
* Receipt of an investigation agent within the past 4 weeks (or within 5 half lives) prior to study initiation
* Systemic corticosteroid therapy within the past month Concurrent use of drugs listed in Appendix C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-10-04 (Actual); Study Completion 2016-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ginette Okoye, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Dept. of Dermatology, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Narrow-band Ultraviolet B Phototherapy | no Intervention
Started | 2 | 0
Completed | 0 | 0
Not Completed | 2 | 0
Not completed — Transportation issues | 1 | 0
Not completed — No enrollment and staff unavailability | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Narrow-band Ultraviolet B Phototherapy | no Intervention | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Vitiligo Area Scoring Index (VASI)
Description: VASI scores of treated versus untreated symmetrical body sites.The percentage of vitiligo involvement is calculated in terms of hand units. One hand unit is approximately equivalent to 1% of the total body surface area. The degree of pigmentation is estimated to the nearest of one of the following percentages: 100% - complete depigmentation, no pigment is present; 90% - specks of pigment present; 75% - depigmented area exceeds the pigmented area; 50% - pigmented and depigmented areas are equal; 25% - pigmented area exceeds depigmented area; and 10% - only specks of depigmentation present. The VASI for each body region is determined by the product of the area of vitiligo in hand units and the extent of depigmentation within each hand unit measured patch. Total body VASI = S All body sites [Hand Units] ´ [Residual depigmentation].
Time Frame: 24 weeks
Population: No participants' data were analyzed, as no pertinent data for the outcome was obtained due to participants drop-out for personal reasons.
Arm/Group | Narrow-band Ultraviolet B Phototherapy | no Intervention
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Dermatology Life Quality Index (DLQI)
Description: Quality of life assessment
Time Frame: 24 weeks
Population: as for outcome 1
Arm/Group | Narrow-band Ultraviolet B Phototherapy | no Intervention
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Skindex-29 Questionnaire
Description: Quality of life assessment
Time Frame: 24 weeks
Population: as for outcome 1
Arm/Group | Narrow-band Ultraviolet B Phototherapy | no Intervention
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Response Stability Index
Time Frame: 24 weeks
Population: as for outcome 1
Arm/Group | Narrow-band Ultraviolet B Phototherapy | no Intervention
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Number of Participants With Histological Change in Tissue Samples
Time Frame: 24 weeks
Population: as for outcome 1
Arm/Group | Narrow-band Ultraviolet B Phototherapy | no Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Narrow-band Ultraviolet B Phototherapy | no Intervention
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 1/2 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Narrow-band Ultraviolet B Phototherapy (N=2) | no Intervention (N=0)
Redness of the skin area in both axillae (armpit) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The main limitation was the fact that study was a long term one and therefore participants could not keep pace with the visits and follow ups

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No